CLINICAL TRIAL: NCT02220322
Title: Age-related Cognitive Change of Femur
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tomidahama Hospital (Other)
Responsible Party: Principal Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Other Study IDs: IRB TH No 9
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Osteoporosis
Keywords: cortical thickness; age
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Age-related change of femur is not well-known. The investigators investigated the longitudinal changes of femur.

DETAILED DESCRIPTION:
Recently, bisphosphonate-related atypical fracture of femur (AFF) is paid attention in clinicians. Almost all AFFs were occurred in thicker cortical thickness. But age-related change of femur is not well-known.

The main objective of this study is to reveal the age-related change of femur.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis or osteopenia patients who presented to our hospital

Exclusion Criteria:

* Patients without osteoporosis or osteopenia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Osteoporosis or osteopenia patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Age-related change of femur | Up to 12 months
  We investigate radiographic features in patients with osteopenia/opsteoporosis. We investigate bilateral femur radiographs concerning to cortical thickening. We analyze age-related change of femur.
  To determine the age-related change of femur , statistical analyses are performed using Spearman correlation, paired t-test, chi-square test, Fisher's exact test and Mann-Whitney U test. Finally, we conclude the effects of age on femur.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Niimi, PhD, Principal Investigator — Tomidahama Hospital
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan